CLINICAL TRIAL: NCT02358161
Title: Phase I/II Study of LDE225 in Combination With Gemcitabine and Nab-paclitaxel in Patients With Locally Advanced or Metastasized Pancreatic Cancer
Brief Title: Phase I/II Study of LDE225 With Gemcitabine and Nab-paclitaxel in Patients With Pancreatic Cancer
Acronym: MATRIX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Novartis (Industry); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, J.W. Wilmink, M.D., PhD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCMEDONC 2013-215; 2013-002370-51 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2015-02-06 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; LDE225; Gemcitabine; nab paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDE225 (Experimental): DLT adn MTD of LED225 co-administered with fixed doses of gemcitabine and nab-paclitaxel in patients with advanced or metastasized pancreatic cancer.
  Interventions: Drug: gemcitabine and nab paclitaxel

INTERVENTIONS:
Drug: gemcitabine and nab paclitaxel — DLT adn MTD of LED225 co-administered with fixed doses of gemcitabine and nab-paclitaxel in patients with advanced or metastasized pancreatic cancer
  Other Names: Gemzar; Abraxane

SUMMARY:
The 5 year survival of patients with locally advanced or metastatic pancreatic cancer is less than 5 %. Since the introduction of gemcitabine, further advances in therapy in the advanced/metastatic setting have been extremely slow. Numerous phase III studies have evaluated different gemcitabine-based regimens as first-line therapy, but in most cases, any observed benefits have been small and restricted to patients with a good performance status (PS). Recently two new chemotherapy combination schedules, FOLFIRINOX and Gemcitabine + nab-paclitaxel demonstrated a significant survival improvement compared to gemcitabine alone. Nab-paclitaxel is especially interesting because it is able to break-down the tumor matrix and increases the concentration of cytotoxic drugs in the tumor.

Our study will explore the modification of the desmoplastic reaction seen in pancreatic cancer using two approaches, targeting tumor stroma by nab-paclitaxel and the hedgehog inhibitor LDE225 and targeting the tumor cells with gemcitabine and nab-paclitaxel.

DETAILED DESCRIPTION:
Growing body of evidence suggests that the stroma is not only a mechanical barrier that may prevent efficient delivery of various anticancer therapies to the tumor, but also constitutes a dynamic compartment of pancreatic tumors that is critically involved in tumor formation, progression and metastasis. Thus, targeting both tumor stroma and cancer cells could be a lucrative strategy to increase the efficacy of our therapeutic approach.

In the present study we want to explore the safety and activity of the chemotherapy combination: Gemcitabine + nab-paclitaxel + LDE225. LDE225 is a hedgehog inhibitor with promising antitumor activity in several cancer models, including pancreatic cancer. One of the main activities is also the degradation of the tumor matrix.

Patients with locally advanced or metastatic pancreatic cancer will be treated with fixed doses of gemcitabine + nab-paclitaxel, the same doses used in the recently presented phase III study (von Hoff American Society of Clinical Oncology ASCO 2013). In the phase I part of the study LDE225 will be added according to standard dose escalation strategy for phase I studies, and at the maximum tolerated dose (MTD) patients will be treated in the phase II part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent according to International Conference on Harmonisation of technical requirements for registration og pharmaceuticals for human use (ICH)/Good cClinical Practice (GCP), and national/local regulations prior to any screening procedures.
2. Male or female adult patients (> 18 years)
3. Patients with histologically/cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma.
4. a. Phase I: patients with non resectable or metastasized pancreatic ductal adenocarcinoma.

   b. Phase II: patients with non resectable or metastasized pancreatic ductal adenocarcinoma not pre-treated with chemotherapy or radiotherapy, unless adjuvant treatment with gemcitabine > 6 months prior to inclusion.
5. Measurable disease as assessed by RECIST 1.1 (Response Evaluation Criteria In Solid Tumors) .
6. ECOG (Eastern Cooperative Oncology Group) (WHO) performance status 0-2
7. Patient has adequate bone marrow and organ function . Patient is able to swallow and retain oral medication

9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;

Exclusion Criteria:

1. History of hypersensitivity to LDE225, or to drugs of similar chemical classes.
2. Patient has received previous treatment with smoothened inhibitors.
3. Patients with known CNS (Central Nervous System) metastases or a primary CNS malignancy.
4. Patients who have neuromuscular disorders or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA (3-hydroxy-3-methyl-glutaryl Coenzyme A) inhibitors (statins), clofibrate and gemfibrozil.
5. Patients who are planning on embarking on new physical activities, such as strenuous exercise, that can result in significant increases in plasma CK (Creatine Kinase) levels while on study treatment.
6. Patients who require the use of coumarin derivates cannot be enrolled as LDE225 is a competitive inhibitors of CYP2C9 based on in-vitro data.
7. Patients with chronic use of corticosteroids
8. Patients who are not willing to avoid consumption of Seville oranges, grapefruit or grapefruit juice grapefruit hybrids, pomelos and exotic citrus fruits during the entire study and preferably 7 days before the first dose of study medications, due to potential CYP3A4 interaction with the study medications.
9. Patients who are not willing to stop taking herbal medications at least 7 days prior to the first dose of study treatment.
10. Patient is currently being treated with drugs known to be strong inhibitors or inducers of CYP3A4/5, which cannot be discontinued or switched to a different medication 7 days prior to starting study treatment and for the duration of the study..
11. Current medical history of the following:

    * History of or presence of clinically significant uncontrolled ventricular or atrial tachyarrhythmia
    * Clinically significant resting bradycardia (< 45 beats per minute) or any primary of secondary heart block
    * History of unstable angina pectoris
    * Clinically significant cardio-vascular disease (e.g. congestive heart failure NYHA Class III-IV (New York Heart Association), atherosclerosis, labile hypertension or uncontrolled hypertension
12. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive HCG (Human Chorionic Gonadotropin) laboratory test
13. Patients who are not willing to apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment.
14. Sexually active males who are unwilling to use a condom during intercourse while taking drug and for 6 months after stopping investigational medications and agree not to father a child in this period. Patients who in the investigators' opinion may be unwilling, unable or unlikely to comply with requirements of the study protocol
15. Patient is currently receiving increasing or chronic treatment with corticosteroids ((≥ the anti-inflammatory potency of 4mg dexamethasone) or another immunosuppressive agent.
16. Patient has been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated before enrollment, may be continued
17. Patient who has received targeted therapy or immunotherapy ≤ 3 weeks (6 weeks for monoclonal antibodies) prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy
18. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LDE225 (e.g., ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
19. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate patient participation in the clinical study.
20. HIV-positive patients on combination antiretroviral therapy.
21. Patients who in the investigators' opinion may be unwilling, unable or unlikely to comply with requirements of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting Toxicity (DLT) and MTD of LDE225 co-administered with gemcitabine and nab-paclitaxel | first six weeks after start treatment
  Phase I: DLT and MTD of LDE225 co-administered with fixed doses of gemcitabine and nab-paclitaxel in patients with advanced or metastasized pancreatic cancer

SECONDARY OUTCOMES:
Median survival | 1 year
Progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: J. W. Wilmink, MD, PhD, Principal Investigator — Academic Medical Center, Medical Oncology
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands